CLINICAL TRIAL: NCT07226141
Title: Valproate for the Treatment of Residual Amblyopia
Acronym: VARA
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Eric Gaier, Assistant Professor of Ophthalmology, Boston Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-P00051999
Record Dates: First submitted 2025-09-26; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-09

CONDITIONS: Amblyopia; Amblyopia Unilateral; Amblyopia, Anisometropic; Amblyopia Strabismic
Keywords: Amblyopia; valproate; valproic acid; pediatric; lazy eye; Histone deacetylase Inhibitor; HDAC; patching; eye patch; visual acuity; visual impairment; critical period; children; ophthalmology
MeSH Terms: conditions — Amblyopia; Vision Disorders | interventions — Valproic Acid; Transdermal Patch

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, double-blind, placebo-controlled interventional study with a cross-over-like design. Participants (ages 8-17) are randomized 1:1 to receive either valproate plus patching followed by placebo plus patching, or placebo plus patching followed by valproate plus patching. Each phase lasts 8 weeks (16 weeks total). The model ensures all participants are exposed to valproate, increases efficiency in a small pilot sample, and allows assessment of durability of response after discontinuation. Randomization is stratified by amblyopia severity, and both participants and investigators are masked to treatment assignment.
Who Masked: Participant, Investigator
Masking Description: Participants, caregivers, investigators, and study staff conducting outcome assessments are all masked to treatment assignment. Study medication (valproate or placebo) is dispensed in identical-appearing capsules and bottles prepared by the research pharmacy. Randomization is managed via a secure web-based system, and treatment codes are not accessible to investigators or participants. Unmasking may only occur in the event of a medical emergency when knowledge of the treatment assignment is essential for subject safety.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 - Placebo first (Placebo Comparator): Participants randomized to Arm 1 will receive oral placebo (250 mg twice daily) in combination with 2 hours of prescribed daily patching for 8 weeks. At the 8-week visit, participants will cross over to oral valproate at an initial dose of 15 mg/kg/day divided twice daily, while continuing the prescribed 2 hours of daily patching for an additional 8 weeks. Dose escalation of valproate up to 30 mg/kg/day (or placebo to 500 mg mice daily) will be permitted at interim visits if visual acuity has not improved and no adverse effects are present. All study medication will be discontinued after 16 weeks, with patching also discontinued at that time.
  Interventions: Drug: Valproate; Drug: Placebo; Behavioral: Patch
- Arm 2 - Valproate first (Experimental): Participants randomized to Arm 2 will receive oral valproate at an initial dose of 15 mg/kg/day divided twice daily, together with 2 hours of prescribed daily patching for 8 weeks. At the 8-week visit, participants will cross over to oral placebo (250 mg twice daily) while continuing 2 hours of daily patching for an additional 8 weeks. If visual acuity has not improved at interim visits and no adverse effects are observed, the valproate dose may be escalated up to 30 mg/kg/day during the initial treatment phase, or placebo increased to 500 mg twice daily during the cross-over phase. After 16 weeks, both study medication and patching will be discontinued.
  Interventions: Drug: Valproate; Drug: Placebo; Behavioral: Patch

INTERVENTIONS:
Drug: Valproate — Valproate is an anti-epileptic medication used in this study to treat amblyopia. Participants will receive valproate in oral tablet form. The dosage will be determined based on the participant's weight and age, following standard dosing guidelines for valproate. The medication will be administered daily for a duration of 8 weeks. Participants will be monitored for any adverse effects, and dosage adjustments will be made if necessary to ensure safety and tolerability.
Drug: Placebo — The placebo intervention consists of an inert substance designed to mimic the appearance and administration of valproate tablets. Participants in the placebo group will receive the placebo tablets daily for the same duration of 8 weeks. This control group will help to assess the efficacy of valproate by comparing outcomes between the valproate and placebo groups. Participants receiving the placebo will also be monitored for any adverse effects to ensure the study's integrity and participant safety.
Behavioral: Patch — Patching is a standard treatment for amblyopia, involving the occlusion of the fellow eye to stimulate the amblyopic eye. Participants will be required to patch their fellow eye for 2 hours daily throughout the 16-week study period. The patching regimen aims to improve visual acuity in the amblyopic eye by encouraging its use. Compliance with the patching protocol will be monitored, and participants will be provided with instructions and support to ensure proper application and adherence to the treatment.

SUMMARY:
The goal of this clinical trial is to determine the efficacy of valproate as an adjunct therapy to treat amblyopia beyond the critical period in children aged 8-17 years who have amblyopia of ≥3 lines of interocular best-corrected (with glasses) visual acuity difference.

The main questions it aims to answer are:

* Does valproate enable clinically meaningful and durable visual recovery from amblyopia?
* Do valproate-treated patients show a change in amblyopic eye visual acuity (lines)? Participants will undergo daily patching for 2 hours (standard of care) plus the addition of valproate or placebo for a total of 16 weeks.

DETAILED DESCRIPTION:
This pilot randomized, double-blind, placebo-controlled clinical trial is designed to evaluate the efficacy and safety of valproate as an adjunctive therapy for residual amblyopia in children and adolescents aged 8-17 years. Amblyopia, the leading cause of monocular visual impairment in children, is responsive to early interventions such as patching and pharmacologic penalization; however, many patients remain with residual visual deficits despite treatment. Current approaches are limited by age-dependent declines in cortical plasticity after closure of the visual system's "critical period."

Valproate (valproic acid), a widely used antiepileptic and mood-stabilizing agent, is also a histone deacetylase (HDAC) inhibitor that promotes synaptic plasticity through chromatin remodeling. Preclinical studies in rodents have demonstrated that HDAC inhibition with valproate restores ocular dominance plasticity and enables recovery of visual function even in adulthood. Translational work has further shown that valproate can reopen critical periods in humans, as evidenced by acquisition of absolute pitch in adult subjects. Together, these data provide strong proof-of-concept support for repurposing valproate as a treatment for amblyopia by reactivating plasticity mechanisms rather than targeting neuromodulatory pathways alone.

In this study, 28 subjects with residual amblyopia (best-corrected amblyopic eye visual acuity 20/40-20/400, stable over ≥8 weeks) will be randomized 1:1 to receive either oral valproate (15 mg/kg/day, divided BID) plus two hours of prescribed daily patching, or oral placebo plus patching, for 8 weeks. After the initial phase, subjects will cross over to the alternate treatment arm for an additional 8 weeks. This cross-over-like design ensures all participants receive valproate, allows assessment of treatment durability, and has precedent in both amblyopia and valproate neuroplasticity studies. Dose escalation up to 30 mg/kg/day will be permitted at interim visits if insufficient visual improvement is observed without adverse effects.

The primary endpoint is change in visual acuity in the amblyopic eye after 8 weeks of treatment. Secondary endpoints include the proportion of patients achieving resolution of amblyopia, change in stereoacuity, durability of treatment response after cross-over, visual acuity in the fellow eye, and prospective evaluation of the valproate safety profile in this population.

Subjects will be monitored closely through a structured schedule of phone calls and in-person visits over 16 weeks. Safety assessments include symptom surveys, liver function tests, complete blood counts, and pregnancy testing as indicated. Standardized visual acuity and stereoacuity testing will be performed at each visit. Compliance will be tracked using patient logs, capsule counts, and investigator assessments.

Potential risks include known adverse effects of valproate, ranging from common but generally mild gastrointestinal and neurological symptoms to rare severe outcomes such as hepatotoxicity, pancreatitis, teratogenicity, and hematologic abnormalities. Subjects will be carefully screened for contraindications, including liver disease, mitochondrial disorders, and pregnancy risk. A Data and Safety Monitoring Committee will oversee adverse event reporting and trial safety.

This trial is intended as a proof-of-concept study to establish feasibility, safety, and preliminary efficacy of valproate for residual amblyopia. Results will inform the design of a larger multicenter randomized trial and provide essential data on effect size, tolerability, and durability of response. If successful, this work could represent a paradigm shift in amblyopia treatment by introducing an epigenetic, plasticity-enhancing approach with the potential for durable recovery of vision in older children and adolescents who currently have limited therapeutic options.

ELIGIBILITY:
Inclusion Criteria:

1. Age 8-17 years
2. Amblyopia associated with strabismus and/or anisometropia

   * Criteria for strabismus: must meet at least one of the following:

     * Heterotropia at distance and/or near with or without spectacle correction
     * History of strabismus surgery
     * Documented history of strabismus that is no longer present and felt by the investigator could have caused the amblyopia
   * Criteria for anisometropia: must meet at least one of the following:

     * ≥ 0.50 D difference in spherical equivalent between eyes
     * ≥ 1.50 D difference in astigmatism in any meridian between the eyes
3. Visual acuity measured in each eye within 7 days prior to enrollment using ETDRS protocol on a study certified visual acuity tester as follows:

   * Amblyopic eye visual acuity of 20/40 - 20/400
   * Sound eye acuity of ≥ 20/25.
4. Current amblyopia treatment (other than spectacle correction)

   * Subjects actively patching at the time of enrollment screening should continue patching through enrollment
   * Visual acuity in amblyopic eye has not improved ≥ 1 line (5 letters) by the same testing method from a previous visit ≥ 8 weeks earlier while on treatment

     * Since this determination is a pre-study examination, the method of visual acuity testing is not mandated
   * Atropine treatment at any time during this pre-enrollment period is not allowed
   * Any treatment prior to the current patching episode with stable acuity is allowed
5. Spectacle correction for measurement of enrollment visual acuity must meet the following criteria and be based on a cycloplegic refraction < 6 months old:

   • Requirement for spectacle correction:
   * Spherical equivalent must be within 0.50 D of fully correcting anisometropia
   * Hyperopia ≥ 3.00 D must be corrected
   * Hyperopia may not be undercorrected by > 1.50 D spherical equivalent and must be symmetrically reduced in each eye
   * Cylinder power must be within 0.50 D of fully correcting the astigmatism
   * Cylinder axis must be within 6 degrees of the axis in the spectacles when the cylinder power is ≥ 1.00 D
   * Myopia of the amblyopic eye > 0.50 D spherical equivalent must be corrected

     ◊ Myopia may not be undercorrected by > 0.25 D or overcorrected by > 0.50D

     • Spectacles meeting the above criteria must be worn:
   * Until visual acuity in amblyopic eye has not improved ≥ 1 line (5 letters) by the same testing method during 2 consecutive visual acuity measurements at least 4 weeks apart (i.e. minimum of 8 weeks spectacle correction) ◊ Since this determination is a pre-study examination, the method of visual acuity testing is not mandated
6. Eye examination within 6 months prior to enrollment
7. Subject must be available for at least 6 months of follow-up, have access to a phone, and be willing to be contacted by clinical staff
8. By investigator judgment, the subject is likely to comply with prescribed treatment (i.e. no prior history of poor compliance with patching) and unlikely to continue to improve with 2 hours of daily patching alone

2.2.2 Exclusions

1. Myopia > -6.00 D spherical equivalent
2. Presence of associated findings that could cause reduced visual acuity

   • Nystagmus does not exclude the subject if the above visual acuity criteria are met
3. Previous intraocular or refractive surgery
4. Strabismus surgery planned within 16 weeks
5. Current vision therapy or orthoptics
6. Known past or present liver or kidney disease
7. Known past or present mitochondrial/metabolic disorder
8. Known past or present psychological problems
9. Known allergies or contraindications to the use of valproate or anti-epileptic medication
10. Current use of medication for the treatment of seizures, bipolar disorder, or migraine, or any medication on the appended list of medications that interact with valproate/valproate acid and its derivatives which can be found here.
11. Prior valproate use
12. Known skin reaction to patch or bandage adhesives
13. Treatment with topical atropine within the past 12 weeks
14. Individuals capable of pregnancy who are pregnant, lactating, or may become pregnant within the next 6 months

    * A negative urine pregnancy test will be required for all participants who have experienced menarche at the time of enrollment
    * Individuals capable of pregnancy must convey an active suitable plan to avoid pregnancy that includes at least one of the following:
    * Hormonal Contraceptives:

      * Combined oral contraceptives (the pill)
      * Contraceptive patch
      * Vaginal contraceptive ring
      * Progestin-only pills
      * Hormonal injections (e.g., Depo-Provera)
      * Hormonal implants (e.g., Nexplanon)
    * Intrauterine Devices (IUDs):

      * Copper IUD (e.g., ParaGard)
      * Hormonal IUDs (e.g., Mirena, Skyla, Liletta)
    * Barrier Methods with Spermicide (less commonly used alone but may be used in combination with other methods for added protection):

      * Male condoms
      * Female condoms
      * Diaphragms with spermicide
      * Cervical caps with spermicide
    * Sterilization:

      * Tubal ligation (for females)
      * Vasectomy (Having a partner who has undergone a vasectomy, confirmed by semen analysis)
    * Abstinence or True Sexual Abstinence:

      o Refraining from heterosexual intercourse
    * Requirements regarding the establishment of pregnancy status and monitoring for pregnancy over the course of the study may be further defined by the IRB

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Amblyopic Eye Best-Corrected Visual Acuity (BCVA) | The comparison will be made between the randomized groups at the 8-week visit, prior to cross-over.
  Change in visual acuity of the amblyopic eye after 8 weeks of treatment with valproate plus patching versus placebo plus patching.

SECONDARY OUTCOMES:
Proportion of patients with resolved amblyopia | 8 weeks
  Proportion of participants achieving resolution of amblyopia, defined as visual acuity in the amblyopic eye of 20/25 or better, following 8 weeks of treatment.
Durability of amblyopic eye visual acuity response | 8 weeks
  Among those in the study arm receiving valproate followed by placebo, the visual acuity in the amblyopic eye will be compared between the 8 week visit (when valproate is discontinued) to the 16 week visit (after completion of placebo). This difference reflects the maintenance of visual acuity and will be analyzed and interpreted in the context of change at an individual level in response to valproate between weeks 0 and 8. The proportion of subjects from the valproate then placebo group maintaining a ≥ 10 letters (2 lines) improvement in the amblyopic eye visual acuity will be calculated and a 95% confidence interval on overall change will be computed.
Change in stereoacuity | 8 weeks and 16 weeks
  Change in log arcsec in stereoacuity assessed with the Randot Preschool Stereoacuity Test. The change in log arcseconds will be compared between groups. Aggregated results will inform how overall stereoacuity has changed, and the difference from baseline will be compared across treatment groups and timepoints.
Quality of life measures using the Pediatric Eye Questionnaire (PedEyeQ) | Change from baseline at 8 weeks and 16 weeks.
  This measure assesses the quality of life deficits across four domains: functional vision, bothered by eyes/vision, social, and frustration/worry. It uses a 3-point frequency scale and Rasch-calibrated domain scores (0-100).
Tolerability and Safety of Valproate | Assessed throughout the study duration at 1,2, 4, 6, 8, 9, 10, 12, 14 and 16 weeks.
  This measure evaluates the tolerability and safety of valproate, assessing the proportion of patients reporting mild, moderate, and severe adverse events, and comparing the proportion of participants requiring dose tapering or de-escalation.

CONTACTS AND LOCATIONS:
Overall Officials: Eric D Gaier, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Waltham, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share individual participant data (IPD) with qualified researchers to promote transparency and further research. Data will be de-identified to ensure privacy and confidentiality. Researchers must submit a formal request outlining their study purpose and intended use of the data. Requests will be reviewed by our study team for ethical and scientific alignment.
  Data will be shared through a secure online repository, accessible to approved researchers. Shared data will include demographic information, clinical outcomes, visual acuity measurements, stereoacuity results, quality of life assessments, and adverse event reports. Researchers must agree to use the data solely for approved purposes and not share it with third parties without consent.
  Researchers are encouraged to publish their findings in peer-reviewed journals and acknowledge the original study and investigators.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The individual participant data (IPD) and supporting information will be available to qualified researchers starting 6 months after the publication of the primary study results. The data will remain accessible for 5 years from the start date. Researchers must submit a formal request, which will be reviewed for ethical and scientific alignment. This plan ensures valuable data contributes to advancements in amblyopia treatment while maintaining confidentiality.
Access Criteria: Who Will Be Able to Access:
  Qualified researchers from academic institutions, research organizations, and healthcare institutions will be able to access the IPD and supporting information. Access will be granted based on the submission and approval of a formal request.
  What They Will Be Able to Access:
  Researchers will have access to de-identified individual participant data, including:
  Demographic information Clinical outcomes Visual acuity measurements Stereoacuity results Quality of life assessments Adverse event reports
  How They Will Be Able to Access:
  Researchers must submit a formal request detailing their study purpose and intended use of the data. The request will be reviewed by our study team for ethical and scientific alignment. Approved researchers will be granted access to the data through a secure online repository that complies with data protection regulations. Access will be restricted to the approved research purposes, and data sharing with third parties will require

REFERENCES:
- [Background] Stewart CE, Fielder AR, Stephens DA, Moseley MJ. Treatment of unilateral amblyopia: factors influencing visual outcome. Invest Ophthalmol Vis Sci. 2005 Sep;46(9):3152-60. doi: 10.1167/iovs.05-0357. PMID 16123414
- [Background] Woodruff G, Hiscox F, Thompson JR, Smith LK. Factors affecting the outcome of children treated for amblyopia. Eye (Lond). 1994;8 ( Pt 6):627-31. doi: 10.1038/eye.1994.157. PMID 7867817
- [Background] Holmes JM, Levi DM. Treatment of amblyopia as a function of age. Vis Neurosci. 2018 Jan;35:E015. doi: 10.1017/S0952523817000220. PMID 29905125
- [Background] Ashrafi MR, Shabanian R, Zamani GR, Mahfelati F. Sodium Valproate versus Propranolol in paediatric migraine prophylaxis. Eur J Paediatr Neurol. 2005;9(5):333-8. doi: 10.1016/j.ejpn.2005.05.004. Epub 2005 Aug 24. PMID 16120482
- [Background] Mattson RH, Cramer JA, Williamson PD, Novelly RA. Valproic acid in epilepsy: clinical and pharmacological effects. Ann Neurol. 1978 Jan;3(1):20-5. doi: 10.1002/ana.410030105. PMID 350128
- [Background] Tomson T, Marson A, Boon P, Canevini MP, Covanis A, Gaily E, Kalviainen R, Trinka E. Valproate in the treatment of epilepsy in girls and women of childbearing potential. Epilepsia. 2015 Jul;56(7):1006-19. doi: 10.1111/epi.13021. Epub 2015 May 16. PMID 25851171
- [Background] Hiilesmaa VK, Bardy AH, Granstrom ML, Teramo KA. Valproic acid during pregnancy. Lancet. 1980 Apr 19;1(8173):883. doi: 10.1016/s0140-6736(80)91387-2. No abstract available. PMID 6103246
- [Background] Nau H, Hauck RS, Ehlers K. Valproic acid-induced neural tube defects in mouse and human: aspects of chirality, alternative drug development, pharmacokinetics and possible mechanisms. Pharmacol Toxicol. 1991 Nov;69(5):310-21. doi: 10.1111/j.1600-0773.1991.tb01303.x. PMID 1803343
- [Background] Cotariu D, Zaidman JL. Developmental toxicity of valproic acid. Life Sci. 1991;48(14):1341-50. doi: 10.1016/0024-3205(91)90430-j. PMID 2008152
- [Background] Shoshany TN, Michalak S, Staffa SJ, Chinn RN, Bishop K, Hunter DG. Effect of Primary Occlusion Therapy in Asymmetric, Bilateral Amblyopia. Am J Ophthalmol. 2020 Mar;211:87-93. doi: 10.1016/j.ajo.2019.10.030. Epub 2019 Nov 9. PMID 31712066
- [Background] Chinn RN, Wilkinson CL, Staffa SJ, Michalak SM, Shoshany TN, Bishop K, Hunter DG, Gaier ED. Amblyopia treatment outcomes in patients with neurodevelopmental disorders. J AAPOS. 2023 Oct;27(5):276.e1-276.e8. doi: 10.1016/j.jaapos.2023.07.014. Epub 2023 Sep 21. PMID 37739211
- [Background] Morrison DG, Heidary G, Chang MY, Binenbaum G, Cavuoto KM, Galvin J, Trivedi R, Kim SJ, Pineles SL. Levodopa/Carbidopa to Augment the Treatment of Amblyopia: A Report by the American Academy of Ophthalmology. Ophthalmology. 2023 Nov;130(11):1221-1227. doi: 10.1016/j.ophtha.2023.07.008. Epub 2023 Aug 29. PMID 37642618
- [Background] Sharif MH, Talebnejad MR, Rastegar K, Khalili MR, Nowroozzadeh MH. Oral fluoxetine in the management of amblyopic patients aged between 10 and 40 years old: a randomized clinical trial. Eye (Lond). 2019 Jul;33(7):1060-1067. doi: 10.1038/s41433-019-0360-z. Epub 2019 Feb 19. PMID 30783259
- [Background] Huttunen HJ, Palva JM, Lindberg L, Palva S, Saarela V, Karvonen E, Latvala ML, Liinamaa J, Booms S, Castren E, Uusitalo H. Fluoxetine does not enhance the effect of perceptual learning on visual function in adults with amblyopia. Sci Rep. 2018 Aug 27;8(1):12830. doi: 10.1038/s41598-018-31169-z. PMID 30150750
- [Background] Chung STL, Li RW, Silver MA, Levi DM. Donepezil Does Not Enhance Perceptual Learning in Adults with Amblyopia: A Pilot Study. Front Neurosci. 2017 Aug 7;11:448. doi: 10.3389/fnins.2017.00448. eCollection 2017. PMID 28824369
- [Background] Wu C, Gaier ED, Nihalani BR, Whitecross S, Hensch TK, Hunter DG. Durable recovery from amblyopia with donepezil. Sci Rep. 2023 Jun 22;13(1):10161. doi: 10.1038/s41598-023-34891-5. PMID 37349338
- [Background] Procianoy E, Fuchs FD, Procianoy L, Procianoy F. The effect of increasing doses of levodopa on children with strabismic amblyopia. J AAPOS. 1999 Dec;3(6):337-40. doi: 10.1016/s1091-8531(99)70041-8. PMID 10613576
- [Background] Mohan K, Dhankar V, Sharma A. Visual acuities after levodopa administration in amblyopia. J Pediatr Ophthalmol Strabismus. 2001 Mar-Apr;38(2):62-7; quiz 96-7. doi: 10.3928/0191-3913-20010301-05. PMID 11310708
- [Background] Leguire LE, Walson PD, Rogers GL, Bremer DL, McGregor ML. Levodopa/carbidopa treatment for amblyopia in older children. J Pediatr Ophthalmol Strabismus. 1995 May-Jun;32(3):143-51. doi: 10.3928/0191-3913-19950501-05. PMID 7636693
- [Background] Leguire LE, Walson PD, Rogers GL, Bremer DL, McGregor ML. Longitudinal study of levodopa/carbidopa for childhood amblyopia. J Pediatr Ophthalmol Strabismus. 1993 Nov-Dec;30(6):354-60. doi: 10.3928/0191-3913-19931101-04. PMID 8120739
- [Background] Leguire LE, Rogers GL, Walson PD, Bremer DL, McGregor ML. Occlusion and levodopa-carbidopa treatment for childhood amblyopia. J AAPOS. 1998 Oct;2(5):257-64. doi: 10.1016/s1091-8531(98)90080-5. PMID 10646745
- [Background] Chatzistefanou KI, Mills MD. The role of drug treatment in children with strabismus and amblyopia. Paediatr Drugs. 2000 Mar-Apr;2(2):91-100. doi: 10.2165/00148581-200002020-00002. PMID 10937461
- [Background] Yang EJ, Lin EW, Hensch TK. Critical period for acoustic preference in mice. Proc Natl Acad Sci U S A. 2012 Oct 16;109 Suppl 2(Suppl 2):17213-20. doi: 10.1073/pnas.1200705109. Epub 2012 Oct 8. PMID 23045690
- [Background] Gervain J, Vines BW, Chen LM, Seo RJ, Hensch TK, Werker JF, Young AH. Valproate reopens critical-period learning of absolute pitch. Front Syst Neurosci. 2013 Dec 3;7:102. doi: 10.3389/fnsys.2013.00102. eCollection 2013. PMID 24348349
- [Background] Lennartsson A, Arner E, Fagiolini M, Saxena A, Andersson R, Takahashi H, Noro Y, Sng J, Sandelin A, Hensch TK, Carninci P. Remodeling of retrotransposon elements during epigenetic induction of adult visual cortical plasticity by HDAC inhibitors. Epigenetics Chromatin. 2015 Dec 14;8:55. doi: 10.1186/s13072-015-0043-3. eCollection 2015. PMID 26673794
- [Background] Shmal D, Mantero G, Floss T, Benfenati F, Maya-Vetencourt JF. Restoring vision in adult amblyopia by enhancing plasticity through deletion of the transcriptional repressor REST. iScience. 2024 Mar 14;27(4):109507. doi: 10.1016/j.isci.2024.109507. eCollection 2024 Apr 19. PMID 38591011
- [Background] Silingardi D, Scali M, Belluomini G, Pizzorusso T. Epigenetic treatments of adult rats promote recovery from visual acuity deficits induced by long-term monocular deprivation. Eur J Neurosci. 2010 Jun;31(12):2185-92. doi: 10.1111/j.1460-9568.2010.07261.x. Epub 2010 Jun 14. PMID 20550570
- [Background] Putignano E, Lonetti G, Cancedda L, Ratto G, Costa M, Maffei L, Pizzorusso T. Developmental downregulation of histone posttranslational modifications regulates visual cortical plasticity. Neuron. 2007 Mar 1;53(5):747-59. doi: 10.1016/j.neuron.2007.02.007. PMID 17329213
- [Background] Monti B, Polazzi E, Contestabile A. Biochemical, molecular and epigenetic mechanisms of valproic acid neuroprotection. Curr Mol Pharmacol. 2009 Jan;2(1):95-109. doi: 10.2174/1874467210902010095. PMID 20021450
- [Background] Penney J, Tsai LH. Histone deacetylases in memory and cognition. Sci Signal. 2014 Dec 9;7(355):re12. doi: 10.1126/scisignal.aaa0069. PMID 25492968
- [Background] Gaier ED, Hunter DG. Advances in Amblyopia Treatment: Paradigm Shifts and Future Directions. Int Ophthalmol Clin. 2017 Fall;57(4):117-128. doi: 10.1097/IIO.0000000000000184. No abstract available. PMID 28885251
- [Background] Falcone MM, Hunter DG, Gaier ED. Emerging therapies for amblyopia. Semin Ophthalmol. 2021 May 19;36(4):282-288. doi: 10.1080/08820538.2021.1893765. Epub 2021 Mar 3. PMID 33656963
- [Background] Holmes JM, Beck RW, Kraker RT, Astle WF, Birch EE, Cole SR, Cotter SA, Donahue S, Everett DF, Hertle RW, Keech RV, Paysse E, Quinn GF, Repka MX, Scheiman MM; Pediatric Eye Disease Investigator Group. Risk of amblyopia recurrence after cessation of treatment. J AAPOS. 2004 Oct;8(5):420-8. doi: 10.1016/S1091853104001612. PMID 15492733
- [Background] Bhola R, Keech RV, Kutschke P, Pfeifer W, Scott WE. Recurrence of amblyopia after occlusion therapy. Ophthalmology. 2006 Nov;113(11):2097-100. doi: 10.1016/j.ophtha.2006.04.034. PMID 17074568
- [Background] Kelly KR, Jost RM, Wang YZ, Dao L, Beauchamp CL, Leffler JN, Birch EE. Improved Binocular Outcomes Following Binocular Treatment for Childhood Amblyopia. Invest Ophthalmol Vis Sci. 2018 Mar 1;59(3):1221-1228. doi: 10.1167/iovs.17-23235. PMID 29625442
- [Background] Giaschi D, Chapman C, Meier K, Narasimhan S, Regan D. The effect of occlusion therapy on motion perception deficits in amblyopia. Vision Res. 2015 Sep;114:122-34. doi: 10.1016/j.visres.2015.05.015. Epub 2015 Jun 4. PMID 26049038
- [Background] Stewart CE, Moseley MJ, Georgiou P, Fielder AR. Occlusion dose monitoring in amblyopia therapy: status, insights, and future directions. J AAPOS. 2017 Oct;21(5):402-406. doi: 10.1016/j.jaapos.2017.06.018. Epub 2017 Sep 7. PMID 28890077
- [Background] Repka MX, Wallace DK, Beck RW, Kraker RT, Birch EE, Cotter SA, Donahue S, Everett DF, Hertle RW, Holmes JM, Quinn GE, Scheiman MM, Weakley DR; Pediatric Eye Disease Investigator Group. Two-year follow-up of a 6-month randomized trial of atropine vs patching for treatment of moderate amblyopia in children. Arch Ophthalmol. 2005 Feb;123(2):149-57. doi: 10.1001/archopht.123.2.149. PMID 15710809
- [Background] Wallace DK; Pediatric Eye Disease Investigator Group; Edwards AR, Cotter SA, Beck RW, Arnold RW, Astle WF, Barnhardt CN, Birch EE, Donahue SP, Everett DF, Felius J, Holmes JM, Kraker RT, Melia M, Repka MX, Sala NA, Silbert DI, Weise KK. A randomized trial to evaluate 2 hours of daily patching for strabismic and anisometropic amblyopia in children. Ophthalmology. 2006 Jun;113(6):904-12. doi: 10.1016/j.ophtha.2006.01.069. PMID 16751033
- [Background] Holmes JM, Lazar EL, Melia BM, Astle WF, Dagi LR, Donahue SP, Frazier MG, Hertle RW, Repka MX, Quinn GE, Weise KK; Pediatric Eye Disease Investigator Group. Effect of age on response to amblyopia treatment in children. Arch Ophthalmol. 2011 Nov;129(11):1451-7. doi: 10.1001/archophthalmol.2011.179. Epub 2011 Jul 11. PMID 21746970
- [Background] Stewart CE, Moseley MJ, Stephens DA, Fielder AR. Treatment dose-response in amblyopia therapy: the Monitored Occlusion Treatment of Amblyopia Study (MOTAS). Invest Ophthalmol Vis Sci. 2004 Sep;45(9):3048-54. doi: 10.1167/iovs.04-0250. PMID 15326120
- [Background] Pediatric Eye Disease Investigator Group Writing Committee; Rutstein RP, Quinn GE, Lazar EL, Beck RW, Bonsall DJ, Cotter SA, Crouch ER, Holmes JM, Hoover DL, Leske DA, Lorenzana IJ, Repka MX, Suh DW. A randomized trial comparing Bangerter filters and patching for the treatment of moderate amblyopia in children. Ophthalmology. 2010 May;117(5):998-1004.e6. doi: 10.1016/j.ophtha.2009.10.014. Epub 2010 Feb 16. PMID 20163869
- [Background] Holmes JM, Kraker RT, Beck RW, Birch EE, Cotter SA, Everett DF, Hertle RW, Quinn GE, Repka MX, Scheiman MM, Wallace DK; Pediatric Eye Disease Investigator Group. A randomized trial of prescribed patching regimens for treatment of severe amblyopia in children. Ophthalmology. 2003 Nov;110(11):2075-87. doi: 10.1016/j.ophtha.2003.08.001. PMID 14597512
- [Background] Repka MX, Beck RW, Holmes JM, Birch EE, Chandler DL, Cotter SA, Hertle RW, Kraker RT, Moke PS, Quinn GE, Scheiman MM; Pediatric Eye Disease Investigator Group. A randomized trial of patching regimens for treatment of moderate amblyopia in children. Arch Ophthalmol. 2003 May;121(5):603-11. doi: 10.1001/archopht.121.5.603. PMID 12742836
- [Background] Pediatric Eye Disease Investigator Group.. A randomized trial of atropine vs. patching for treatment of moderate amblyopia in children. Arch Ophthalmol. 2002 Mar;120(3):268-78. doi: 10.1001/archopht.120.3.268. PMID 11879129
- [Background] Hatt SR, Leske DA, Castaneda YS, Wernimont SM, Liebermann L, Cheng-Patel CS, Birch EE, Holmes JM. Understanding the Impact of Residual Amblyopia on Functional Vision and Eye-related Quality of Life Using the PedEyeQ. Am J Ophthalmol. 2020 Oct;218:173-181. doi: 10.1016/j.ajo.2020.05.039. Epub 2020 Jun 5. PMID 32511967
- [Background] Gonzalez EG, Wong AM, Niechwiej-Szwedo E, Tarita-Nistor L, Steinbach MJ. Eye position stability in amblyopia and in normal binocular vision. Invest Ophthalmol Vis Sci. 2012 Aug 9;53(9):5386-94. doi: 10.1167/iovs.12-9941. PMID 22789926
- [Background] Chung ST, Kumar G, Li RW, Levi DM. Characteristics of fixational eye movements in amblyopia: Limitations on fixation stability and acuity? Vision Res. 2015 Sep;114:87-99. doi: 10.1016/j.visres.2015.01.016. Epub 2015 Feb 7. PMID 25668775
- [Background] Subramanian V, Jost RM, Birch EE. A quantitative study of fixation stability in amblyopia. Invest Ophthalmol Vis Sci. 2013 Mar 19;54(3):1998-2003. doi: 10.1167/iovs.12-11054. PMID 23372053
- [Background] Birch EE, Kelly KR, Giaschi DE. Fellow Eye Deficits in Amblyopia. J Binocul Vis Ocul Motil. 2019 Jul-Sep;69(3):116-125. doi: 10.1080/2576117X.2019.1624440. Epub 2019 Jun 4. PMID 31161888
- [Background] Birch EE, Jost RM, Wang YZ, Kelly KR, Giaschi DE. Impaired Fellow Eye Motion Perception and Abnormal Binocular Function. Invest Ophthalmol Vis Sci. 2019 Aug 1;60(10):3374-3380. doi: 10.1167/iovs.19-26885. PMID 31387113
- [Background] Kelly KR, Cheng-Patel CS, Jost RM, Wang YZ, Birch EE. Fixation instability during binocular viewing in anisometropic and strabismic children. Exp Eye Res. 2019 Jun;183:29-37. doi: 10.1016/j.exer.2018.07.013. Epub 2018 Jul 10. PMID 30006273
- [Background] McKee SP, Levi DM, Movshon JA. The pattern of visual deficits in amblyopia. J Vis. 2003;3(5):380-405. doi: 10.1167/3.5.5. PMID 12875634
- [Background] Birch EE. Amblyopia and binocular vision. Prog Retin Eye Res. 2013 Mar;33:67-84. doi: 10.1016/j.preteyeres.2012.11.001. Epub 2012 Nov 29. PMID 23201436